CLINICAL TRIAL: NCT03855215
Title: Implementation of CRP Point of Care Testing in Primary Care to Improve Antibiotic Targeting in Respiratory Illness (ICAT)
Acronym: ICAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oxford University Clinical Research Unit, Vietnam (Other)
Collaborators: National Hospital for Tropical Diseases, Hanoi, Vietnam (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 31HN
Record Dates: First submitted 2019-02-11; First posted 2019-02-26 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Acute Respiratory Infection
Keywords: acute respiratory infection; ARI; antibiotic; Antimicrobial resistance; AMR; primary health care; CRP

STUDY DESIGN:
Intervention Model Description: The implementation of CRP point of care tests will be conducted at commune health centres (CHCs), the primary access point for public health services in Vietnam (CHC details are described in the Location section below). Prior to introduction of the tests, an educational session will be provided for local healthcare workers in both intervention and control arms about the role of antibiotics and AMR. After randomization, further training will be provided for healthcare workers in the intervention CHCs as to the use of CRP testing to guide antibiotic prescribing decisions. In the intervention CHCs, healthcare workers will be trained on the use and interpretation of CRP testing in ARI (detailed in section 5.4). Educational materials will also be developed for patients and care-givers regarding the value of CRP testing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The ACTIM CRP Rapid Test (Medix, Biochemica) will be made available to the healthcare workers at the CHCs for use in patients in the target population.
  Printed guidance will be issued for the performance and interpretation of the CRP test results in terms of antibiotic guided treatment. The treating healthcare worker will decide based on their clinical evaluation whether or not to comply with this guideline. This guidance will also be discussed during the training sessions.
  The healthcare workers are recommended to use the CRP tests in all patients meeting the target population. The CRP cut-offs will be recommended below in the absence of warning signs of severity:
  CRP level < 10 mg/L: no antibiotics are recommended CRP level from 10 mg/L to 40 mg/L: antibiotics are unlikely to be needed but should be considered in cases of high clinical concern CRP level > 40 mg/L: antibiotics are recommended.
  Interventions: Diagnostic Test: ACTIM CRP Rapid Test (Medix, Biochemica)
- Control (No Intervention): Working as routine

INTERVENTIONS:
Diagnostic Test: ACTIM CRP Rapid Test (Medix, Biochemica) — The implementation of CRP point of care tests will be conducted at commune health centres (CHCs), the primary access point for public health services in Vietnam. In the intervention CHCs, healthcare workers will be trained on the use and interpretation of CRP testing in ARI. healthcare workers can decide to follow the test results or not.
  Arms: Intervention

SUMMARY:
The proposed study will monitor and evaluate a quality improvement project - the introduction of commercially available lateral flow CRP tests with international regulatory approval, as a routine care service to improve the management of patients with acute respiratory infection (ARI) and reduce unnecessary antibiotic prescribing. No research staff will be present, and to minimise disruption and alteration of routine care, a waiver of written patient informed consent will be requested from the relevant ethical review boards, in accordance with the 2016 WHO/CIOMS International Guidance for Health-related Research Involving Humans8. Instead, patients in intervention clusters will be provided with information concerning how the test can assist healthcare workers in identifying when antibiotics are required, after which they will be free to refuse its use.

The test selected for use in the study is the Actim® CRP test from Medix Biochemica (Finland; ISO certification ISO13485:2016). The test is a simple lateral flow device that uses capillary blood, obtained through a finger/heel puncture. The test provides a semi-quantitative indication of whether CRP concentrations are <10mg/L, between 10-40mg/L, between 40-80mg/L, or above 80mg/L, in under 5 minutes with minimal training requirements. The test has been approved by the European regulatory body (CE-marking) as well as in 13 other countries around the world (including Switzerland, Norway, Iceland, Israel and Thailand) and has been validated for accuracy in previous publications.9,10 Our own research group has also confirmed the tests' accuracy in both laboratory and field environments, including their thermos-stability in a tropical climate (see annex). Neither Medix Biochemica nor any of its distributors, have had involvement with the design of the evaluation and our group has no conflict of interest with respect to the choice of the test.

Main research question: Can point of care CRP tests introduced in routine primary healthcare reduce prescription of antibiotics for patients with acute respiratory infections, outside of the research context?

Brief description of the intervention: The implementation of CRP point of care tests will be conducted at commune health centres (CHCs), the primary access point for public health services in Vietnam (CHC details are described in the Location section below). Prior to introduction of the tests, an educational session will be provided for local healthcare workers in both intervention and control arms about the role of antibiotics and AMR. After randomization, further training will be provided for healthcare workers in the intervention CHCs as to the use of CRP testing to guide antibiotic prescribing decisions. In the intervention CHCs, healthcare workers will be trained on the use and interpretation of CRP testing in ARI (detailed in section 5.4). Educational materials will also be developed for patients and care-givers regarding the value of CRP testing.

Description of the population to be studied: This study will be conducted in the general population of Nam Dinh, a rural province in northern Vietnam. The test will be provided at CHCs and recommended for use in patients presenting with a chief complaint of ARI.

DETAILED DESCRIPTION:
STUDY PROCEDURES

1. Screening and Recruitment - A list of potential CHCs will be compiled by province-level officials, and those meeting eligibility criteria will be invited to take part. CHCs will be randomly allocated to intervention or routine care arms using a computer-generated random allocation procedure.

   If baseline variability in antibiotic prescribing practices is identified from reviewing retrospective routine records, high and low prescription centres will be stratified.

   In the intervention CHCs, patients with ARIs will be provided leaflets with information about CRP testing, antibiotics and AMR. Healthcare workers will then decide whether to use a CRP test as part of routine care of patients with ARI. Patients' autonomy will be respected and as with any medical procedure this test can be declined. In the control CHCs patients will be provided with an information leaflet regarding the need for rational use of antibiotics in ARIs but with no mention of CRP testing.
2. Clinical assessment - All patients will have a medical history taken and will be examined as per normal practice. In the control arm, local guidelines and WHO IMCI recommendations will guide treatment. In the intervention arm, doctors can choose to use CRP test results in addition to existing guidelines.
3. General training and education - Healthcare worker training - Before the study sites (CHCs) are randomized, an overview of the study will be presented to all local healthcare workers and provide education about the role of antibiotics, antimicrobial resistance and identification of clinical signs of severity as well as good clinical practice (GCP) for research.

   Patient education - Educational materials will be developed for patients and care-givers regarding antibiotic use and AMR. These will be available to patients presenting with ARIs in both arms, with additional information regarding the CRP tests added to the intervention group leaflets.
4. Intervention - CRP test - The ACTIM CRP Rapid Test (Medix, Biochemica) will be made available to the healthcare workers at the CHCs for use in patients in the target population.

   Printed guidance will be issued for the performance and interpretation of the CRP test results in terms of antibiotic guided treatment. The treating healthcare worker will decide based on their clinical evaluation whether or not to comply with this guideline. This guidance will also be discussed during the training sessions.

   As the purpose of the study is to establish whether antibiotic prescription rates can be reduced by using CRP POC test results, the healthcare workers are recommended to use the CRP tests in all patients meeting the target population. The CRP cut-offs below are recommended in the absence of warning signs of severity:

   CRP level < 10 mg/L: no antibiotics are recommended CRP level from 10mg/L to 40 mg/L: antibiotics are unlikely to be needed but should be considered in cases of high clinical concern CRP level > 40 mg/L: antibiotics are recommended. Based on the previous clinical trial of CRP testing in ARI in Vietnam in similar CHCs, it's anticipated approximately 75% of patients to have CRP levels below 10mg/L, 20% between 10-40mg/L and 5% above 40 mg/L6.

   Healthcare worker training - Additional training will be provided to healthcare workers in the intervention arm. Findings from previous CRP studies have been used to inform the training and guidance for the healthcare workers.

   Face-to-face training will be provided on how the test could be used to inform their prescribing behaviour and a practical session on CRP testing. Content will include which patients should be offered CRP tests; CRP cut-off values; safety nets and caution in result interpretation (including danger signs from IMCI13 and IMAI14 guidelines and patients with co-morbidities). Healthcare workers will be advised that the CRP cut offs are guidelines and that antibiotics can be prescribed or withheld according to their clinical judgement. If the healthcare worker feels the patient requires referral to a higher level facility this should be done without delay and that the CRP tests should not be used in these cases. The training will be provided by the study team in the local language.

   The CHCs and healthcare workers will be given a telephone number to contact should any queries arise during the study. Laminated posters and desk reminders with the CRP cut-off values will be given to the intervention sites.In addition to general information about rational antibiotic use contained in the patient leaflet, patients in the intervention arm will have an extra section explaining the role of CRP testing to guide antibiotic prescriptions.

   Patient education - Patients with ARIs in all CHCs will be provided with an information leaflet regarding rational use of antibiotics in ARI and the implications of overuse of antibiotics for the development of AMR. An additional section for the intervention arm will explain the role of CRP testing to guide antibiotic prescriptions.
5. Clinical/laboratory/other procedures - CRP tests will be available for healthcare workers to use in ARI patients consulting at intervention CHCs. If patient agree to take the test, a finger prick blood sample will be taken by the CHC staff and placed on a semi-quantitative lateral flow CRP test-kit (Actim® CRP, Medix Biochemica, Finland). Results will be available within 5-10 minutes. Other than the finger prick sample for the CRP test no samples will be taken or stored. CRP test kits and other consumables will be re-stocked on a monthly basis provided and checked to confirm they are properly used for study the study purposes only.
6. Withdrawal of participants from the study - Healthcare workers will be free to refrain from using the tests and they are not obliged to follow the guidelines in their antibiotic prescribing. Healthcare workers will also be free to decline the interviews on the usability and acceptability of the tests. Patients' autonomy will be respected and they will be free to decline the CRP test.
7. Minimization of Error and Bias - To reduce bias within healthcare providers, cluster randomisation will be used so that the same doctors will not see patients in both the intervention and control groups. The study will be conducted for 1 year to allow for seasonal variation. To measure outcomes, electronic patient record data captured routinely in health station log books will be used. This information is a requirement for national health insurance reimbursements, and will be captured in the same way in each arm. Health-workers in both arms will receive data quality training at the start of the study period.
8. Serious adverse events monitoring - As the research poses no more than minimal risks to participants, a data and safety monitory board (DSMB) will not be required. Based on previous studies it's anticipated that no serious adverse events associated with the CRP tests and patients will not be followed up. However, data on admissions for ARI at hospitals serving this catchment population will be retrospectively requested. Health insurance numbers will be used to link with primary healthcare records, in order to identify any study patients who were subsequently hospitalised. This will be done at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 1 to under 65 years old
* First consultation with an acute respiratory infection diagnosed by the healthcare worker with at least 1 focal sign or symptom*
* Symptoms lasting less than 7 days * Focal signs and symptoms: (1) cough, (2) rhinitis (sneezing, nasal congestion, or runny nose), (3) pharyngitis (sore throat), (4) shortness of breath, (5) wheezing, (6) chest pain, or (7) auscultation abnormalities.

Exclusion Criteria:

* Patients requiring referral to a higher level facility based on the healthcare worker's clinical assessment
* immunosuppressed patients (known HIV, long term steroid use)
* those with a suspicion of tuberculosis or a non-respiratory tract illness

Ages: 1 Year to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2606 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients aged 1 to 65 years, consulting for ARI, who are prescribed antibiotics in the two study arms | Through study completion, the proportion of 1 year

SECONDARY OUTCOMES:
The proportion of patients that consulted with ARI in the preceding year. | Before the 1st recruitment
Prescription rates for ARI patients in the preceding year. | Before the 1st recruitment
Proportion of patients indicated CRP test according to diagnosis, age, gender | Through study completion, the data of 1 year
Proportion of patients prescribed an antibiotic in the intervention arm with: a. CRP < 10 mg/L b. CRP from 10mg/L to 40mg/L c. CRP > 40mg/L | Through study completion, the proportion of 1 year
Proportion of patients receiving an antibiotic with the denominator being: a. All attendances b. All non-routine attendances | Through study completion, the proportion of 1 year
Proportion of patients receiving an antibiotic prescription by diagnosis, age, season, recorded fever, sex | Through study completion, the proportion of 1 year
The proportion of patients referred to a higher level facility at the initial consultation by checking the e-database of health insurance (HI) reimbursement | Through study completion, the proportion of 1 year
Proportion of patients in whom the test is indicated who re-attend the health facility within a 30 days period, and whether antibiotics were prescribed comparing intervention CHCs and controls | Through study completion, the proportion of 1 year
Proportion of patients in whom the test is indicated hospitalised within a 30 day period (excluding patients referred at consultation) | 30 days after the last recruitment
Qualitatively measure the usability and acceptability of CRP test among healthcare workers | After finishing the recruitment, organize the structured interviews, ask about 1 year of study implementation
  Structured interviews will be conducted with the healthcare workers in both the intervention and control arms at the end of the study for their views on antibiotic use and AMR. Healthcare workers in the intervention arm will also be asked whether the test was usable and useful and whether they support their continued use
Measure of cost-effectiveness | Through study completion, estimate the cost-effectiveness of the intervention for 1 year
  A cost analysis will be carried out to assess the budget implications for introducing the tests, accounting for the cost of treatments and referrals, and a cost-benefit analysis will compare any incremental costs with the modelled costs of AMR averted
the proportion of patients in whom use of the test was recommended that received the test. | Through study completion, the proportion of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- National Hospital for Tropical Diseases, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaya Z, Kucukcongar A, Vuralli D, Emeksiz HC, Gursel T. Leukocyte populations and C-reactive protein as predictors of bacterial infections in febrile outpatient children. Turk J Haematol. 2014 Mar;31(1):49-55. doi: 10.4274/Tjh.2013.0057. Epub 2014 Mar 5. PMID 24764729
- [Background] Goossens H, Ferech M, Vander Stichele R, Elseviers M; ESAC Project Group. Outpatient antibiotic use in Europe and association with resistance: a cross-national database study. Lancet. 2005 Feb 12-18;365(9459):579-87. doi: 10.1016/S0140-6736(05)17907-0. PMID 15708101
- [Background] Shallcross LJ, Davies DS. Antibiotic overuse: a key driver of antimicrobial resistance. Br J Gen Pract. 2014 Dec;64(629):604-5. doi: 10.3399/bjgp14X682561. No abstract available. PMID 25452508
- [Background] Greer RC, Intralawan D, Mukaka M, Wannapinij P, Day NPJ, Nedsuwan S, Lubell Y. Retrospective review of the management of acute infections and the indications for antibiotic prescription in primary care in northern Thailand. BMJ Open. 2018 Jul 30;8(7):e022250. doi: 10.1136/bmjopen-2018-022250. PMID 30061442
- [Background] Aabenhus R, Jensen JU, Jorgensen KJ, Hrobjartsson A, Bjerrum L. Biomarkers as point-of-care tests to guide prescription of antibiotics in patients with acute respiratory infections in primary care. Cochrane Database Syst Rev. 2014 Nov 6;(11):CD010130. doi: 10.1002/14651858.CD010130.pub2. PMID 25374293
- [Background] Do NT, Ta NT, Tran NT, Than HM, Vu BT, Hoang LB, van Doorn HR, Vu DT, Cals JW, Chandna A, Lubell Y, Nadjm B, Thwaites G, Wolbers M, Nguyen KV, Wertheim HF. Point-of-care C-reactive protein testing to reduce inappropriate use of antibiotics for non-severe acute respiratory infections in Vietnamese primary health care: a randomised controlled trial. Lancet Glob Health. 2016 Sep;4(9):e633-41. doi: 10.1016/S2214-109X(16)30142-5. Epub 2016 Aug 3. PMID 27495137
- [Background] Althaus T, Greer RC, Swe MMM, Cohen J, Tun NN, Heaton J, Nedsuwan S, Intralawan D, Sumpradit N, Dittrich S, Doran Z, Waithira N, Thu HM, Win H, Thaipadungpanit J, Srilohasin P, Mukaka M, Smit PW, Charoenboon EN, Haenssgen MJ, Wangrangsimakul T, Blacksell S, Limmathurotsakul D, Day N, Smithuis F, Lubell Y. Effect of point-of-care C-reactive protein testing on antibiotic prescription in febrile patients attending primary care in Thailand and Myanmar: an open-label, randomised, controlled trial. Lancet Glob Health. 2019 Jan;7(1):e119-e131. doi: 10.1016/S2214-109X(18)30444-3. PMID 30554748
- [Background] Evrard B, Roszyk L, Fattal S, Dastugue B, Sapin V. [Evaluation of rapid, semi-quantitative assay of C-reactive protein in whole blood, Actim CRP]. Ann Biol Clin (Paris). 2005 Sep-Oct;63(5):525-9. French. PMID 16230290
- [Background] Brouwer N, van Pelt J. Validation and evaluation of eight commercially available point of care CRP methods. Clin Chim Acta. 2015 Jan 15;439:195-201. doi: 10.1016/j.cca.2014.10.028. Epub 2014 Oct 31. PMID 25445415
- [Background] Senn N, Rarau P, Salib M, Manong D, Siba P, Rogerson S, Mueller I, Genton B. Use of antibiotics within the IMCI guidelines in outpatient settings in Papua New Guinean children: an observational and effectiveness study. PLoS One. 2014 Mar 13;9(3):e90990. doi: 10.1371/journal.pone.0090990. eCollection 2014. PMID 24626194
- [Background] WHO. Integrated Management of Childhood Illness. Geneva, Switzerland; 2014
- [Background] The World Health Organization. Integrated management of adolescent and adult illness: interim guidelines for first-level facility health workers at health centre and district outpatient clinic: acute care. 2009; Rev 3
- [Background] Sim J, Dawson A. Informed consent and cluster-randomized trials. Am J Public Health. 2012 Mar;102(3):480-5. doi: 10.2105/AJPH.2011.300389. Epub 2012 Jan 19. PMID 22390511
- [Background] Lubell Y, Blacksell SD, Dunachie S, Tanganuchitcharnchai A, Althaus T, Watthanaworawit W, Paris DH, Mayxay M, Peto TJ, Dondorp AM, White NJ, Day NP, Nosten F, Newton PN, Turner P. Performance of C-reactive protein and procalcitonin to distinguish viral from bacterial and malarial causes of fever in Southeast Asia. BMC Infect Dis. 2015 Nov 11;15:511. doi: 10.1186/s12879-015-1272-6. PMID 26558692
- [Derived] Do NTT, Vu TVD, Greer RC, Dittrich S, Vandendorpe M, Pham NT, Ta DN, Cao HT, Khuong TV, Le TBT, Duong TH, Nguyen TH, Cai NTH, Nguyen TQT, Trinh ST, van Doorn HR, Lubell Y, Lewycka S. Implementation of point-of-care testing of C-reactive protein concentrations to improve antibiotic targeting in respiratory illness in Vietnamese primary care: a pragmatic cluster-randomised controlled trial. Lancet Infect Dis. 2023 Sep;23(9):1085-1094. doi: 10.1016/S1473-3099(23)00125-1. Epub 2023 May 22. PMID 37230105
- [Derived] Thi Thuy Do N, Greer RC, Lubell Y, Dittrich S, Vandendorpe M, Nguyen VA, Ngoc Thach P, Thi Dieu Ngan T, Van Kinh N, Hung Thai C, Dung LTK, Nguyen Thi Cam T, Nguyen TH, Nadjm B, van Doorn HR, Lewycka S. Implementation of C-reactive protein point of care testing to improve antibiotic targeting in respiratory illness in Vietnamese primary care (ICAT): a study protocol for a cluster randomised controlled trial. BMJ Open. 2020 Dec 23;10(12):e040977. doi: 10.1136/bmjopen-2020-040977. PMID 33361164
- See also: Ministry of Health. Vietnam health service delivery profile — http://www.wpro.who.int/health_services/service_delivery_profile_vietnam.pdf
- See also: World Health Organisation. International ethical guidelines for health-related research involving humans. — https://cioms.ch/wp-content/uploads/2017/01/WEB-CIOMS-EthicalGuidelines.pdf